CLINICAL TRIAL: NCT03706521
Title: A Phase 2, 52 Week, Single Center, Open-Label Study Utilizing Imaging Techniques and Evaluating the Safety and Efficacy of SM04690 Injectable Suspension for the Treatment of Moderately to Severely Symptomatic Knee Osteoarthritis
Brief Title: A Study Utilizing Imaging Techniques and Evaluating the Safety and Efficacy of SM04690 for the Treatment of Moderately to Severely Symptomatic Knee Osteoarthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to COVID-19-related issues.
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM04690-OA-08
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Knee Osteoarthritis
Keywords: SM04690; Wnt pathway inhibitor; osteoarthritis; Samumed; lorecivivint; Biosplice Therapeutics, Inc.
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — lorecivivint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 0.07 mg SM04690 (Experimental): Single intra-articular injection of 0.07 mg SM04690 in 2 mL vehicle
  Interventions: Drug: SM04690

INTERVENTIONS:
Drug: SM04690 — Healthcare professional-administered intra-articular injection performed once on Day 1 of the study.
  Other Names: lorecivivint

SUMMARY:
This phase 2 study is a single center, open-label study of SM04690 injected intraarticularly (IA) into the target knee (most painful) joint of moderately to severely symptomatic osteoarthritis (OA) subjects at a single dose of 0.07 mg SM04690 per 2 mL injection. This study will utilize magnetic resonance imaging (MRI) (including T1rho and T2 mapping pulse sequence MRI, three-dimensional spoiled gradient recalled [3D-SPGR] pulse sequence MRI, and whole organ MRI scoring [WORMS]), radiographic imaging, Western Ontario and McMaster Universities Arthritis Index (WOMAC) and patient reported outcomes (PROs) for data collection to assess efficacy outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory (single assistive devices such as canes allowed if needed less than 50% of the time, subjects requiring a walker are excluded)
* Diagnosis of femorotibial OA in the target knee by standard American College of Rheumatology (ACR) criteria at the Screening Visit (clinical AND radiographic criteria); OA of the knee is not to be secondary to any rheumatologic conditions (e.g., rheumatoid arthritis)
* Pain compatible with OA of the knee(s) for at least 26 weeks prior to the Screening Visit
* Primary source of pain throughout the body is due to OA in the target knee
* Daily OA knee pain diary average Numeric Rating Scale (NRS) intensity score ≥4 and ≤8 in the target knee on the 11-point (0-10) NRS scale for the 7 days immediately preceding Day 1
* Pain NRS scores recorded for the target knee on at least 4 out of the 7 days immediately preceding Day 1
* Daily OA knee pain diary average NRS intensity score <4 in the non-target knee on the 11-point (0-10) NRS scale for the 7 days immediately preceding Day 1
* Pain NRS scores recorded for the non-target knee on at least 4 out of the 7 days immediately preceding Day 1
* Baseline mJSW by radiograph between 2 and 4 mm, inclusive, in the target knee at the Screening Visit as assessed by independent central readers
* Total WOMAC score of 96-192 (out of 240) for the target knee at Day 1 regardless of if the subject is on symptomatic oral treatment
* Negative drug test for amphetamine, methamphetamine, buprenorphine, cocaine, methadone, opiates, phencyclidine (PCP), propoxyphene, barbiturates, benzodiazepine, methaqualone, and tricyclic antidepressants, except if any such drugs are clinically indicated and allowed by the protocol at the Screening Visit
* Subjects with depression or anxiety must be clinically stable for 12 weeks prior to the Screening Visit and, if on treatment for depression or anxiety, be on 12 weeks of stable therapy
* Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
* Subjects must have read and understood the informed consent form, and must have signed it prior to any study-related procedure being performed
* Subject's Screening Visit must occur while enrollment into the study is open

Exclusion Criteria:

* Women who are pregnant, lactating, or have a positive pregnancy test result at the Screening Visit
* Women of childbearing potential who are sexually active, and who are not willing to use an acceptable method of birth control during the study period
* Men of childbearing potential who are sexually active and have a partner who is capable of becoming pregnant, neither of whom are agreeable to using an acceptable method of birth control during the study period
* Body mass index (BMI) > 40
* Partial or complete joint replacement in either knee
* Currently requires: a) regular use (in the opinion of the Investigator) of ambulatory assistive devices (e.g., wheelchair, parallel bars, walker, canes, or crutches), or b) use of a lower extremity prosthesis, and/or a structural knee brace (i.e., a knee brace that contains hardware)
* Radiographic disease Stage 0, 1, or 4 in the target knee at the Screening Visit according to the Kellgren-Lawrence (KL) grading of knee OA as assessed by independent central readers
* Previous treatment with SM04690
* Subjects who have previously failed screening on this protocol and fail to meet re-screening criteria
* Any surgery (e.g., arthroscopy) in either knee within 26 weeks prior to the Screening Visit
* Any surgery scheduled during the study period. Non-surgical invasive procedures conducted for a diagnostic or therapeutic purpose scheduled during the study period are not prohibited
* Significant and clinically evident misalignment of either knee that would impact subject function, as determined by the Investigator
* History of malignancy within the last 5 years; however, subjects with prior history of in situ basal or squamous cell skin cancer are eligible if completely excised. Subjects with other malignancies are eligible if they have been continuously disease free for at least 5 years prior to the Screening Visit
* Clinically significant abnormal screening hematology values, blood chemistry values, or urinalysis values as determined by the Investigator
* Any condition, including laboratory findings not included in the Screening Visit laboratory tests and findings in the medical history or in the pre-study assessments, that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
* Comorbid conditions that could affect study endpoint assessments of the target knee, including, but not limited to, rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, gout or pseudogout, and fibromyalgia
* Other conditions that, in the opinion of the Investigator, could affect study endpoint assessments of either knee, including, but not limited to, peripheral neuropathy (e.g., diabetic neuropathy), symptomatic hip osteoarthritis, symptomatic degenerative disc disease, and patellofemoral syndrome
* Any diagnosed psychiatric condition that includes, but is not limited to, a history of mania, bipolar disorder, psychotic disorder, schizophrenia, schizoaffective disorder, major depressive disorder, or generalized anxiety disorder
* Participation in a clinical research trial that included the receipt of an investigational product or any experimental therapeutic procedure, or an observational research trial related to osteoarthritis within 8 weeks prior to to the Screening Visit, or planned participation in any such trial; the last date of participation in the trial, not the last date of receipt of investigational product, must be at least 8 weeks prior to the Screening Visit
* Any intra-articular injection into the target knee with a therapeutic aim including, but not limited to, viscosupplementation (e.g., hyaluronic acid), platelet-rich plasma (PRP), and stem cell therapies within 24 weeks prior to the Screening Visit; treatment of the target knee with intra-articular glucocorticoids greater than 12 weeks prior to the Screening Visit is allowed
* Treatment with systemic glucocorticoids greater than 10 mg prednisone or the equivalent per day within 4 weeks prior to the Screening Visit
* Effusion of the target knee clinically requiring aspiration within 12 weeks prior to the Screening Visit
* Use of electrotherapy, acupuncture, and/or chiropractic treatments for knee OA within 4 weeks prior to the Screening Visit
* Any known active infections, including urinary tract infection, upper respiratory tract infection, sinusitis, suspicion of intra-articular infection, hepatitis B or hepatitis C infection, and/or infections that may compromise the immune system such as human immunodeficiency virus (HIV) at Day 1
* Current use, or use within 12 weeks prior to the Screening Visit, of centrally acting analgesics
* Current use, or use within 12 weeks prior to the Screening Visit, of anticonvulsants (refer to Appendix 2)
* Subjects requiring the usage of opioids >1x per week within 12 weeks prior to the Screening Visit
* Topical local anesthetic agents (gels, creams, or patches such as the Lidoderm patch) used for the treatment of knee OA within 7 days of the Screening Visit
* Any chronic condition that has not been well controlled or subjects with a chronic condition who have not maintained a stable therapeutic regimen of a prescription therapy in the opinion of the investigator. In addition, subjects with an HbA1c >9 at the Screening Visit will be excluded.
* If on nonsteroidal anti-inflammatory drugs (NSAIDs) for the treatment of OA pain, subjects who have not maintained a stable regimen in the opinion of the Investigator at the Screening Visit
* Any contraindications for performing MRI
* Subjects who have a current or pending disability claim, workers' compensation, or litigation(s) that may compromise response to treatment
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at any investigative site, or are directly affiliated with the study at any investigative site
* Subjects employed by Samumed, LLC, or any of its affiliates or development partners (that is, an employee, temporary contract worker, or designee) responsible for the conduct of the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cartilage thickness in the target knee | Baseline and Week 26
  Evaluate change from baseline in cartilage thickness in the target knee as measured by 3D-SPGR pulse sequence MRI
Change from baseline in cartilage volume in the target knee | Baseline and Week 26
  Evaluate change from baseline in cartilage volume in the target knee as measured by 3D-SPGR pulse sequence MRI
Change from baseline in cartilage quality in the target knee | Baseline and Week 26
  Evaluate change from baseline in cartilage quality in the target knee determined by the increase or decrease in proteoglycan and glycosaminoglycan (GAG) content and hydration as measured by T1rho and T2 mapping pulse sequence MRI

SECONDARY OUTCOMES:
Change from baseline in cartilage thickness in the target knee | Baseline, Weeks 13 and 52
  Evaluate change from baseline in cartilage thickness in the target knee as measured by 3D-SPGR pulse sequence MRI
Change from baseline in cartilage volume in the target knee | Baseline, Weeks 13 and 52
  Evaluate change from baseline in cartilage volume in the target knee as measured by 3D-SPGR pulse sequence MRI
Change from baseline in cartilage quality in the target knee | Baseline, Weeks 13 and 52
  Evaluate change from baseline in cartilage quality in the target knee by the increase or decrease in proteoglycan and GAG content and hydration as measured by T1rho and T2 mapping pulse sequence MRI
Change from baseline in total Whole Organ MRI Scoring (WORMS) in the target knee | Baseline, Weeks 13, 26, and 52
  Evaluate change from baseline in total WORMS in the target knee
Change from baseline OA pain in the target knee | Baseline, Weeks 13, 26, and 52
  Evaluate change from baseline OA pain in the target knee as assessed by Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain subscore
Change from baseline OA function in the target knee | Baseline, Weeks 13, 26, and 52
  Evaluate change from baseline OA function in the target knee as assessed by WOMAC physical function subscore
Change from baseline symptoms of OA in the target knee | Baseline, Weeks 13, 26, and 52
  Evaluate change from baseline symptoms of OA in the target knee as assessed by WOMAC total score
Change from baseline OA disease activity | Baseline, Weeks 13, 26, and 52
  Evaluate change from baseline OA disease activity as assessed by Patient Global Assessment
Change from baseline in medial joint space width (mJSW) of the target knee | Baseline, Weeks 26 and 52
  Evaluate change from baseline in mJSW as documented by radiograph of the target knee
Change from baseline in cartilage thickness in the non-target knee | Baseline, Weeks 13, 26, and 52
  Evaluate change from baseline in cartilage thickness in the non-target knee as measured by 3D-SPGR pulse sequence MRI
Change from baseline in cartilage volume in the non-target knee | Baseline, Weeks 13, 26, and 52
  Evaluate change from baseline in cartilage volume in the non-target knee as measured by 3D-SPGR pulse sequence MRI
Change from baseline in cartilage quality in the non-target knee | Baseline, Weeks 13, 26, and 52
  Evaluate change from baseline in cartilage quality in the non-target knee determined by the increase or decrease in proteoglycan and GAG content and hydration as measured by T1rho and T2 mapping pulse sequence MRI
Change from baseline in total WORMS in the non-target knee | Baseline, Weeks 13, 26, and 52
  Evaluate change from baseline in total WORMS in the non-target knee
Change from baseline in mJSW of the non-target knee | Baseline, Weeks 26 and 52
  Evaluate change from baseline in mJSW as documented by radiograph of the non-target knee

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (1):
- Research Site, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No